CLINICAL TRIAL: NCT04347954
Title: Effect of PVP-I Nasal Sprays vs Normal Saline Nasal Sprays on SARS-CoV-2 Nasopharyngeal Titers
Brief Title: PVP-I Nasal Sprays and SARS-CoV-2 Nasopharyngeal Titers (for COVID-19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-56134
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Results first posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: nasal spray; PVP-I; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Povidone-Iodine 2% (Experimental): Participants will administer PVP-I 2% nasal spray for 5 days. Nasopharyngeal swabs will be taken on Day 1 at baseline, Day 1 at four hours post-first dose, and Day 5.
  Participants will complete a daily symptom journal from Day 1 through Day 5.
  Interventions: Drug: Povidone-Iodine 2%
- Povidone-Iodine 0.5% (Experimental): Participants will administer PVP-I 0.5% nasal spray for 5 days. Nasopharyngeal swabs will be taken on Day 1 at baseline, Day 1 at four hours post-first dose, and Day 5.
  Participants will complete a daily symptom journal from Day 1 through Day 5
  Interventions: Drug: Povidone-Iodine 0.5%
- Isotonic saline 0.9% (Placebo Comparator): Participants will administer two sprays of isotonic saline nasal spray for 5 days. Nasopharyngeal swabs will be taken on Day 1 at baseline, Day 1 at four hours post-first dose, and Day 5.
  Participants will complete a daily symptom journal from Day 1 through Day 5.
  Interventions: Drug: Isotonic saline 0.9%

INTERVENTIONS:
Drug: Povidone-Iodine 2% — Two sprays to each nare of PVP-I 2% via nasal spray bottle, four times a day
  Arms: Povidone-Iodine 2%
Drug: Povidone-Iodine 0.5% — Two sprays to each nare of PVP-I 0.5% via nasal spray bottle, four times a day
  Arms: Povidone-Iodine 0.5%
Drug: Isotonic saline 0.9% — Two sprays to each nare of isotonic saline (0.9% NaCl) via nasal spray bottle, four times a day
  Arms: Isotonic saline 0.9%

SUMMARY:
The study aims to determine the safety and efficacy of povidone-iodine (PVP-I) containing nasal sprays as compared to isotonic saline nasal sprays in COVID-19 positive patients. The primary outcome measure is SARS-CoV-2 viral titers in the nasal cavity and nasopharynx. In vitro studies have shown PVP-I to be highly virucidal against the viruses which cause SARS and MERS. Additionally, clinical studies have shown PVP-I saline sprays to be well tolerated in human subjects. PVP-I oral rinses and sprays have been trialed as methods to reduce the incidence and symptoms of viruses which cause the "common cold."

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 by lab test within 5 days of study participation

Exclusion Criteria:

* Allergy to "iodine," shellfish, or food dye
* Receiving intranasal steroids
* Sinus surgery within 30 days of beginning the study
* Intubated at the time of enrollment
* Pregnancy
* Participation in other COVID-19 studies - to be determined on a case by case basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2020-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayakar V. Nayak, MD, PhD, Principal Investigator — Stanford University; Neelaysh Vukkadala, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 265 patients were assessed for eligibility; 47 patients were randomized into the study,
Groups:
- Isotonic Saline 0.9%: Participants administer 2 sprays of isotonic saline (0.9% NaCl) to each nare via nasal spray bottle, four times a day for 5 days.
- Povidone-Iodine 0.5%: Participants administer 2 sprays of povidone-iodine (PVP-I) 0.5% to each nare via nasal spray bottle, four times a day for 5 days.
- Povidone-Iodine 2%: Participants administer 2 sprays of PVP-I 2% to each nare via nasal spray bottle, four times a day for 5 days.
Period: Overall Study
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
Started | 15 | 15 | 17
Received Allocated Intervention | 12 | 15 | 14
Negative PCR Swab at Baseline | 1 | 3 | 1
Completed | 12 | 14 | 14
Not Completed | 3 | 1 | 3
Not completed — Did not present to study site for allocated intervention | 3 | 0 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received the allocated intervention and completed the study; participants with negative PCR nasal swab results at baseline or incomplete data were excluded.
Groups:
- Povidone-Iodine 0.5%: Participants administer 2 sprays of PVP-I 0.5% to each nare via nasal spray bottle, four times a day for 5 days.
- Total: Total of all reporting groups
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2% | Total
Number analyzed (Participants) | 11 | 11 | 13 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (15.6) | 45.2 (12.2) | 40.7 (19.9) | 43.2 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 5 | 18
  Male | 3 | 6 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 7 | 10 | 25
  Hispanic | 1 | 3 | 3 | 7
  Asian | 2 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 13 | 35
Days since positive COVID test to enrollment [Mean (Standard Deviation); unit: days] | 3.9 (2.8) | 3.7 (1.5) | 3.0 (1.1) | 3.5 (1.9)
Days since symptoms to enrollment [Mean (Standard Deviation); unit: days] | 4.8 (2.2) | 7.2 (2.6) | 7.1 (3.2) | 6.3 (2.8)
Active tobacco use [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0
Comorbidities [Count of Participants; unit: Participants]
  Sinusitis/allergy | 2 | 1 | 0 | 3
  Respiratory disease/Asthma | 2 | 0 | 0 | 2
  Cardiac disease | 0 | 1 | 1 | 2
  Neurodegenerative disease | 0 | 0 | 0 | 0
Prior Treatment [Count of Participants; unit: Participants]
  Saline nasal irrigations | 0 | 1 | 0 | 1
  Tylenol/NSAIDs | 0 | 0 | 1 | 1
  None | 11 | 10 | 12 | 33
Noted change to taste or smell at enrollment [Count of Participants; unit: Participants] | 5 | 6 | 8 | 19
Risk factors for smell loss [Count of Participants; unit: Participants]
  History of head trauma | 0 | 0 | 0 | 0
  History of sinus surgery | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Cycle Threshold (Ct) Values Through Day 3 as a Measure of Change in Viral Titers of SARS-CoV-2
Description: Nasopharyngeal swabs were obtained and quantitative reverse transcription-polymerase chain reaction (RT-PCR) testing was performed to determine the viral load in the nasopharynx.
  Cycle threshold (Ct) denotes how many PCR cycles are required before the SARS-CoV-2 viral RNA reached a detectable level. Higher Ct values correspond to lower viral copy numbers. For reference, Ct values of 20 correspond to ~2.12 x 106 viral copies per milliliter, while a Ct value of 40 is undetectable and is considered the lower limit of detection of this RT-PCR test for SARS-CoV-2.
Time Frame: Day 1 (baseline), Day 1 (1 hour), Day 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
Number analyzed (Participants) | 11 | 11 | 13
cycles
  Baseline | 24.36 (6.83) | 26.03 (4.86) | 28.42 (6.42)
  Hour 1 | 25.71 (6.87) | 26.46 (5.36) | 27.45 (8.09)
  Day 3 | 29.20 (6.82) | 36.26 (21.56) | 31.01 (7.12)
Statistical Analysis 1: Comparison: Isotonic Saline 0.9% vs Povidone-Iodine 0.5%; Analysis of change in mean Ct values incorporating baseline, hour 1, and day 3 values; Test type: Other; Mean Difference (Net) = -0.349, 95% CI 2-sided [-1.584 to 0.886]
Statistical Analysis 2: Comparison: Isotonic Saline 0.9% vs Povidone-Iodine 2%; Analysis of change in mean Ct values incorporating baseline, hour 1, and day 3 values; Test type: Other; Mean Difference (Net) = -1.059, 95% CI 2-sided [-2.318 to 0.201]

2. Secondary Outcome: Count of Participants Experiencing Adverse Events of Interest After Nasal Sprays
Description: Participants were asked on day 3 whether they experienced the adverse event since baseline, then asked on day 5 whether they experienced the adverse event since day 3 (collected by questionnaire). Adverse events of interest include: Nasal burning/pain, headaches, ear pain, sneezing, and nose bleeds.
Time Frame: Assessed on days 3 and 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
Number analyzed (Participants) | 11 | 11 | 13
Participants
  Nasal burning or pain - Day 3 | 4 | 2 | 13
  Nasal burning or pain - Day 5 | 2 | 2 | 13
  Headaches - Day 3 | 3 | 3 | 5
  Headaches - Day 5 | 2 | 2 | 6
  Ear pain - Day 3 | 1 | 0 | 2
  Ear pain - Day 5 | 1 | 0 | 2
  Sneezing - Day 3 | 4 | 1 | 9
  Sneezing - Day 5 | 4 | 1 | 9
  Nose bleeds - Day 3 | 1 | 0 | 1
  Nose bleeds - Day 5 | 1 | 0 | 1

3. Secondary Outcome: Count of Participants Experiencing Fevers as a Measure of Frequency of Symptoms Related to SARS-CoV-2
Description: Count of participants that experienced fevers at either mild, moderate, or severe intensity. Participants were asked on day 3 whether they experienced the symptom since baseline, then asked on day 5 whether they experienced the symptom since day 3. Participants rated the severity of their symptoms on a 4-point Likert scale with "1" representing 'not experiencing that symptom,' "2" representing mild symptoms, "3" representing 'moderate symptoms,' and "4" representing 'severe symptoms.'
Time Frame: Assessed on days 3 and 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
Number analyzed (Participants) | 11 | 11 | 13
Participants
  Day 3 - Mild | 0 | 0 | 0
  Day 3 - Moderate | 1 | 0 | 0
  Day 3 - Severe | 0 | 0 | 0
  Day 5 - Mild | 0 | 0 | 0
  Day 5 - Moderate | 0 | 0 | 0
  Day 5 - Severe | 1 | 0 | 0

4. Secondary Outcome: Count of Participants Experiencing Chills as a Measure of Frequency of Symptoms Related to SARS-CoV-2
Description: Count of participants that experienced chills at either mild, moderate, or severe intensity. Participants were asked on day 3 whether they experienced the symptom since baseline, then asked on day 5 whether they experienced the symptom since day 3. Participants rated the severity of their symptoms on a 4-point Likert scale with "1" representing 'not experiencing that symptom,' "2" representing mild symptoms, "3" representing 'moderate symptoms,' and "4" representing 'severe symptoms.'
Time Frame: Assessed on days 3 and 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
Number analyzed (Participants) | 11 | 11 | 13
Participants
  Day 3 - Mild | 1 | 0 | 1
  Day 3 - Moderate | 2 | 0 | 0
  Day 3 - Severe | 0 | 0 | 0
  Day 5 - Mild | 2 | 0 | 0
  Day 5 - Moderate | 1 | 0 | 0
  Day 5 - Severe | 1 | 0 | 0

5. Secondary Outcome: Count of Participants Experiencing Fatigue as a Measure of Frequency of Symptoms Related to SARS-CoV-2
Description: Count of participants that experienced fatigue at either mild, moderate, or severe intensity. Participants were asked on day 3 whether they experienced the symptom since baseline, then asked on day 5 whether they experienced the symptom since day 3. Participants rated the severity of their symptoms on a 4-point Likert scale with "1" representing 'not experiencing that symptom,' "2" representing mild symptoms, "3" representing 'moderate symptoms,' and "4" representing 'severe symptoms.'
Time Frame: Assessed on days 3 and 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
Number analyzed (Participants) | 11 | 11 | 13
Participants
  Day 3 - Mild | 4 | 5 | 6
  Day 3 - Moderate | 1 | 2 | 0
  Day 3 - Severe | 1 | 0 | 0
  Day 5 - Mild | 3 | 3 | 2
  Day 5 - Moderate | 2 | 3 | 0
  Day 5 - Severe | 0 | 0 | 0

6. Secondary Outcome: Count of Participants Experiencing Loss of Sense of Smell as a Measure of Frequency of Symptoms Related to SARS-CoV-2
Description: Count of participants that experienced loss of sense of smell at either mild, moderate, or severe intensity. Participants were asked on day 3 whether they experienced the symptom since baseline, then asked on day 5 whether they experienced the symptom since day 3. Participants rated the severity of their symptoms on a 4-point Likert scale with "1" representing 'not experiencing that symptom,' "2" representing mild symptoms, "3" representing 'moderate symptoms,' and "4" representing 'severe symptoms.'
Time Frame: Assessed on days 3 and 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
Number analyzed (Participants) | 11 | 11 | 13
Participants
  Day 3 - Mild | 2 | 3 | 2
  Day 3 - Moderate | 0 | 2 | 1
  Day 3 - Severe | 2 | 1 | 4
  Day 5 - Mild | 2 | 2 | 3
  Day 5 - Moderate | 1 | 2 | 2
  Day 5 - Severe | 1 | 1 | 1

7. Secondary Outcome: Count of Participants Experiencing Loss of Sense of Taste as a Measure of Frequency of Symptoms Related to SARS-CoV-2
Description: Count of participants that experienced loss of sense of taste at either mild, moderate, or severe intensity. Participants were asked on day 3 whether they experienced the symptom since baseline, then asked on day 5 whether they experienced the symptom since day 3. Participants rated the severity of their symptoms on a 4-point Likert scale with "1" representing 'not experiencing that symptom,' "2" representing mild symptoms, "3" representing 'moderate symptoms,' and "4" representing 'severe symptoms.'
Time Frame: Assessed on days 3 and 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
Number analyzed (Participants) | 11 | 11 | 13
Participants
  Day 3 - Mild | 3 | 4 | 3
  Day 3 - Moderate | 0 | 1 | 0
  Day 3 - Severe | 1 | 1 | 3
  Day 5 - Mild | 0 | 1 | 2
  Day 5 - Moderate | 1 | 2 | 1
  Day 5 - Severe | 0 | 1 | 2

8. Secondary Outcome: Count of Participants Experiencing Nasal Congestion as a Measure of Frequency of Symptoms Related to SARS-CoV-2
Description: Count of participants that experienced nasal congestion at either mild, moderate, or severe intensity. Participants were asked on day 3 whether they experienced the symptom since baseline, then asked on day 5 whether they experienced the symptom since day 3. Participants rated the severity of their symptoms on a 4-point Likert scale with "1" representing 'not experiencing that symptom,' "2" representing mild symptoms, "3" representing 'moderate symptoms,' and "4" representing 'severe symptoms.'
Time Frame: Assessed on days 3 and 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
Number analyzed (Participants) | 11 | 11 | 13
Participants
  Day 3 - Mild | 5 | 5 | 7
  Day 3 - Moderate | 3 | 2 | 4
  Day 3 - Severe | 0 | 0 | 0
  Day 5 - Mild | 5 | 4 | 6
  Day 5 - Moderate | 2 | 1 | 0
  Day 5 - Severe | 0 | 0 | 0

9. Secondary Outcome: Count of Participants Experiencing Sore Throat as a Measure of Frequency of Symptoms Related to SARS-CoV-2
Description: Count of participants that experienced sore throat at either mild, moderate, or severe intensity. Participants were asked on day 3 whether they experienced the symptom since baseline, then asked on day 5 whether they experienced the symptom since day 3. Participants rated the severity of their symptoms on a 4-point Likert scale with "1" representing 'not experiencing that symptom,' "2" representing mild symptoms, "3" representing 'moderate symptoms,' and "4" representing 'severe symptoms.'
Time Frame: Assessed on days 3 and 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
Number analyzed (Participants) | 11 | 11 | 13
Participants
  Day 3 - Mild | 4 | 0 | 4
  Day 3 - Moderate | 0 | 0 | 0
  Day 3 - Severe | 0 | 0 | 0
  Day 5 - Mild | 1 | 0 | 2
  Day 5 - Moderate | 0 | 0 | 0
  Day 5 - Severe | 0 | 0 | 0

10. Secondary Outcome: Compliance With Study Drug Administration
Description: Participants were asked to estimated doses completed at day 5 (0-25%, 26-50%, 51-75%, or 76-100%). The count of participants who estimated their compliance to be within each range is reported.
Time Frame: 5 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
Number analyzed (Participants) | 11 | 11 | 13
Participants
  76-100% compliant | 11 | 11 | 13
  51-75% compliant | 0 | 0 | 0
  26-50% compliant | 0 | 0 | 0
  0-25% compliant | 0 | 0 | 0

11. Secondary Outcome: Count of Participants Normosmia, Microsmia, or Anosmia as a Measure of Change in the University of Pennsylvania Smell Identification Test (UPSIT)
Description: Participants scratch test cards and attempt to identify the smell from a multiple choice set of options. Their scores are then computed and categorized as normosmia (normal), mild, moderate, or severe microsmia (loss of smell), or anosmia (total loss of smell).
Time Frame: Day 1 (baseline), Day 30
Population: Participants who received the allocated intervention and completed the study and with data available for the respective time point; participants with negative PCR nasal swab results at baseline or incomplete data were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
Number analyzed (Participants) | 11 | 11 | 13
Participants
  Anosmia - Baseline: number analyzed (Participants) | 11 | 10 | 12
  Anosmia - Baseline | 2 | 4 | 5
  Anosmia - day 30: number analyzed (Participants) | 10 | 11 | 12
  Anosmia - day 30 | 0 | 0 | 0
  Severe microsmia - baseline: number analyzed (Participants) | 11 | 10 | 12
  Severe microsmia - baseline | 3 | 1 | 1
  Severe microsmia - day 30: number analyzed (Participants) | 10 | 11 | 12
  Severe microsmia - day 30 | 2 | 1 | 1
  Moderate microsmia - baseline: number analyzed (Participants) | 11 | 10 | 12
  Moderate microsmia - baseline | 2 | 2 | 2
  Moderate microsmia - day 30: number analyzed (Participants) | 10 | 11 | 12
  Moderate microsmia - day 30 | 0 | 0 | 1
  Mild microsmia - baseline: number analyzed (Participants) | 11 | 10 | 12
  Mild microsmia - baseline | 2 | 0 | 3
  Mild microsmia - day 30: number analyzed (Participants) | 10 | 11 | 12
  Mild microsmia - day 30 | 5 | 2 | 3
  Normosmia - baseline: number analyzed (Participants) | 11 | 10 | 12
  Normosmia - baseline | 2 | 3 | 1
  Normosmia - day 30: number analyzed (Participants) | 10 | 11 | 12
  Normosmia - day 30 | 3 | 8 | 7

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Isotonic Saline 0.9% | Povidone-Iodine 0.5% | Povidone-Iodine 2%
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 6/15 | 6/15 | 13/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Isotonic Saline 0.9% (N=15) | Povidone-Iodine 0.5% (N=15) | Povidone-Iodine 2% (N=17)
Nasal burning (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 13
Headaches (Nervous system disorders) | 4 | 3 | 7
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 11
Nosebleeds (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2

LIMITATIONS AND CAVEATS:
The study did not meet its accrual goal of 45 participants with analyzable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT04347954/Prot_SAP_000.pdf